CLINICAL TRIAL: NCT04124237
Title: Long Term Monitoring to Detect Risk of Sudden Death in Inherited Arrhythmia Patients
Brief Title: Long Term Monitoring for Risk of Sudden Death
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Kingston Health Sciences Centre (Other); Quebec Heart Institute (Other); Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Andrew Krahn, Professor Department of Medicine University of British Columbia, Chief of Cardiology, University of British Columbia
Other Study IDs: H15-00658
Record Dates: First submitted 2017-03-29; First posted 2019-10-11 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Inherited Cardiac Arrhythmias; Long QT Syndrome; Arrhythmogenic Right Ventricular Cardiomyopathy; Brugada Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia
Keywords: Inherited Heart Rhythms; Genetic Heart Conditions; Sudden Cardiac Arrest; Sudden Cardiac Death
MeSH Terms: conditions — Long QT Syndrome; Arrhythmogenic Right Ventricular Dysplasia; Brugada Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood Samples drawn:
  1 X 9 ml EDTA
  DNA samples for bio banking will be stored long-term
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Risk prediction in in inherited heart rhythm conditions that may cause sudden cardiac arrest or death is difficult. Sometimes the risks may be low but the loss of life in an otherwise healthy young individual is catastrophic. Clinicians often treat to the extreme to prevent this and so often those at unknown risk for a serious cardiac event are treated with an implanted cardioverter defibrillator (ICD) to protect against sudden death even though the risk is low or unknown. ICDs them selves are not without adverse events such as needing battery replacements, mechanical complications, inappropriate shocks and body image and self esteem issues for the patient. This study will use an inject able monitor that is less invasive to monitor inherited heart rhythm patients long term to help gather long term heart rhythm data (3 years) on patients with an inherited heart rhythm that will help to detect symptoms of dangerous heart rhythms so that the appropriate care can be provided.

DETAILED DESCRIPTION:
Risk stratification is challenging in latent genetically mediated sudden death syndromes, where the absolute risks are low but the loss of life is catastrophic in otherwise well young individuals. Countering this is the manifest drawbacks of liberal use of Implantable Cardioverter Defibrillator (ICDs) in this population, who may suffer harm from the limitations of ICDs with respect to repeated generator changes, lead/mechanical complications, non-target shocks and issues with body image and self esteem. This balance is struck with patients and clinicians in the inherited arrhythmia clinics daily.

The Principal Investigator has a longstanding interest in cardiac monitoring and syncope, with extensive experience with cardiac monitoring technologies. Recently published data from the study team indicates that 69% of unexplained cardiac arrest patients had suffered syncope, presyncope, chest pain or palpitations, significantly greater than the 43% incidence in their first-degree relatives8. The prevalence of syncope was 34% in those patients with subsequently diagnosed inherited causes of cardiac arrest. This suggests an excellent opportunity to detect symptomatic and asymptomatic arrhythmias in patients to risk stratify patients and direct ICD resources to patients that are likely to benefit. Coupling of recording with remote monitoring of device-detected events enables a short time from detected arrhythmia to reporting and resultant clinical decision-making (base station in the patient's home transmits any acquired data daily).

An intermediate risk population is seen regularly in the inherited arrhythmia clinic, based on a wide array of clinical features that are proven or suspected risk markers in patients who either prefer to avoid an ICD, or whose risk is insufficient to clearly warrant an ICD. The risk in these individuals is hampered by the relatively uncommon short-term risk of spontaneous arrhythmia that is detected by routine 24-48 Holter surveillance to assist as a "tie breaker", to favor more aggressive therapy with an ICD. This study will extend the monitoring period of intermediate risk patients to 3 years and enable detection of symptomatic and asymptomatic ventricular arrhythmia that would inform risk discussion with the patient and favor more aggressive therapy. The latter may involve incremental drug therapy, cardiac sympathectomy or an ICD.

Loop recorder implantation (Reveal LINQ, Medtronic, Minneapolis MN), also called an insertable cardiac monitor (ICM) has the ability to analyze the beat to beat variability of cardiac cycles on a 2 minute ECG strip and stores the tracing for visual confirmation of any cardiac events. The device also provides the patient with the ability to activate the device manually and so facilitates analysis of heart rhythm during symptomatic events.

The device is manufactured and will be provided by Medtronic Canada Ltd, 99 Hereford Street, Brampton, Ontario L6Y 0R3 +1 905-460-3800. The Medtronic Reveal LINQ is a programmable device that continuously monitors a patient's ECG and other physiological parameters. The device records cardiac information in response to automatically detected arrhythmias and patient activation. The form factor of the device has changed from that similar to a USB thumb drive that requires surgical implantation to that of a paper clip that can be injected in a minimally invasive environment including office based clean rooms. This device is small leadless and is inserted under the skin, in the chest. The device can be inserted by the physician in the office, saving precious healthcare resources.

Potential Adverse Events include but are not limited to:

* Device rejection phenomena (including local tissue reaction)
* Device migration
* Infection
* Erosion through the skin

ELIGIBILITY:
Inclusion Criteria:

1. Inherited Heart Rhythm (IHR) patient with breakthrough symptoms on best medical care that does not warrant an ICD, or patient declines ICD:

   * Syncope or seizure that is suspected to be arrhythmic in nature with a Brugada pattern on ECG
   * Long QT syndrome (LQTS)or Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT) on beta blocker
   * Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) with at least 2 minor or 1 major 2010 task force criteria,

     * must be more than isolated disease causing gene positive
2. Asymptomatic IHR patient with extreme phenotype, does not warrant an ICD

   * spontaneous persistent type 1 Brugada pattern
   * macroscopic T wave alternates on resting ECG, Holter monitor or exercise test (especially Long QTS)
   * QTc > 500 msec in LQTS, other than LQT1
   * persistent asymptomatic bidirectional couplets or non-sustained PMVT in CPVT with exercise on therapy (including beta blocker and flecainide)
   * definite ARVC with some high risk feature (first degree relative with SCD, couplets or nsVT on Holter)
3. Double mutation carrier IAC patient (at least one definite and one probable disease causing)
4. Patient with class 1 indication for ICD who declines it (patient or parent declines, example: young patient with cardiac arrest)
5. High-risk Cardiac arrest survivors with preserved ejection fraction (CASPER) unexplained cardiac arrest (UCA) patients and family members, defined as 2 or more of 1) previous syncope suspected to be arrhythmic 2) exercise recovery QTc ≥455 msec 3) epinephrine 0.10 μg/kg/min Δ QT ≥30 msec 4) Valt>0, k>3during Holter9 5) QTVI >95th %ile (>-1) on Holter9.
6. High-risk patient not otherwise described above presented to an adjudication Committee with ≥75% consensus of risk.
7. Willing signed informed consent form
8. Ages 2 and over may participate (pediatric cases will be considered in Pediatric Centres only after the first 10 pilot cases are completed and reviewed by the DSMB Specialized pediatric procedures will be in developed by the pediatric clinicians)

Exclusion Criteria:

1. Unable or unwilling to give informed consent
2. ICD or pacemaker in place or considered preferable by the treating physician and/or patient/parent.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Risk stratification is challenging in latent genetically mediated sudden death syndromes, where the absolute risks are low but the loss of life is catastrophic in otherwise well young individuals. Countering this is the manifest drawbacks of liberal use of Implantable Cardioverter Defibrillator (ICDs) in this population, who may suffer harm from the limitations of ICDs with respect to repeated generator changes, lead/mechanical complications, non-target shocks and issues with body image and self esteem. This balance is struck with patients and clinicians in the inherited arrhythmia clinics daily.
Sampling Method: Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Detection of ≥5 beats of non-sustained wide QRS complex tachycardia (i.e. likely to be VT). | From time of implant to time of cardiac event requiring intervention (maximum 3 years)
  The number of irregular heart rates requiring change in treatment

SECONDARY OUTCOMES:
Time to diagnosis | From time of implant to time of recorded finding indicating a diagnosis (maximum 3 years)
  Time to determine risk and required intervention
ICD implant rate | From time of implant to time of preventative treatment (maximum 3 years)
  How many participants will require treatment with an implanted cardioverter defibrillator
Mortality | Time of implant until date of death (maximum 3 years)
  In the event of a death the cause will be classified by the site investigator as cardiac, non cardiac, sudden and non sudden
ICM Complication rate | Time of implant to time of treatment for complication (maximum 3 years)
  Number of problems related to the device, infection, pain, premature removal

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krahn, Dr., Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No